CLINICAL TRIAL: NCT06800846
Title: Comparative Analgesic Effect After Total Knee Arthroplasty Between Intraosseous Multimodal Analgesic Agent Injection Versus Periarticular Injection - A Randomized Control Trial
Brief Title: Comparative Analgesic Effect After Total Knee Arthroplasty Between Intraosseous and Peri-articular Injection
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Yot Tanariyakul, Comparative analgesic effect after total knee arthroplasty between intraosseous multimodal analgesic agent injection versus periarticular injection - A Randomized Control Trial, Thammasat University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUH Intraosseous injection TKA
Record Dates: First submitted 2025-01-18; First posted 2025-01-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Pain Postoperative; Total Knee Anthroplasty; Functional Outcomes
Keywords: peri-articular injection; intraosseous injection; multimodal analgesia cocktail; TKA; pain postoperative; functional outcomes
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intraosseous multimodal analgesia injection (Experimental): Participants received combinations of 0.5% bupivacaine 100 mg + 0.1% adrenaline 0.6 mg + Morphine 5mg + Ketorolac 30 mg (totally 22 ml) which divided by 12 ml inject into intramedullary canal before bone plug impaction to close the canal and 10 ml inject into metaphysis of tibia before cementation and implantation
  Interventions: Procedure: Intraosseous Morphine
- peri-articular multimodal analgesia injection (Active Comparator): Participants received combinations of 0.5% bupivacaine 100 mg + 0.1% adrenaline 0.6 mg + Morphine 5mg + Ketorolac 30 mg and mix with normal saline solution for totally 75 ml which divided by 25 ml inject into medial gutter and 25 ml inject into lateral gutter before cementation and implantation. And the last 25 ml of multimodal analgesic drugs were injected into quadriceps.
  Interventions: Procedure: Periarticular Injection

INTERVENTIONS:
Procedure: Intraosseous Morphine — Participants received combinations of 0.5% bupivacaine 100 mg + 0.1% adrenaline 0.6 mg + Morphine 5mg + Ketorolac 30 mg (totally 22 ml) which divided by 12 ml inject into intramedullary canal before bone plug impaction to close the canal and 10 ml inject into metaphysis of tibia before cementation and implantation
  Other Names: intraosseous injection
  Arms: Intraosseous multimodal analgesia injection
Procedure: Periarticular Injection — Participants received combinations of 0.5% bupivacaine 100 mg + 0.1% adrenaline 0.6 mg + Morphine 5mg + Ketorolac 30 mg and mix with normal saline solution for totally 75 ml which divided by 25 ml inject into medial gutter and 25 ml inject into lateral gutter before cementation and implantation. And the last 25 ml of multimodal analgesic drugs were injected into quadriceps.
  Other Names: peri-articular injection
  Arms: peri-articular multimodal analgesia injection

SUMMARY:
The goal of this RCT is to compare analgesic effect after total knee arthroplasty between intraosseous multimodal analgesic agent injection versus periarticular injection. The main question[s] it aims to answer are: Does Intraosseous multimodal analgesic cocktail injection have more post-operative analgesic effect than Peri-articular injection in patients who have done TKA (P)? Participants will randomized to intraosseous injection group or peri-articular injection group and will record the 100-mm VAS pain scores for 2 weeks after TKA. Researchers will compare to peri-articular injection group to see pain and functional outcomes after TKA.

DETAILED DESCRIPTION:
Intra-operatively, you will be randomly assigned to receive intraosseous multimodal analgesic agent injection or peri-articular multimodal analgesic agent injection along with other standard medications. In the intraosseous injection group: Participants received combinations of 0.5% bupivacaine 100 mg + 0.1% adrenaline 0.6 mg + Morphine 5mg + Ketorolac 30 mg (totally 22 ml) which divided by 12 ml inject into intramedullary canal before bone plug impaction to close the canal and 10 ml inject into metaphysis of tibia before cementation and implantation. In the peri-articualr injection group: Participants received combinations of the same drug and mix with normal saline solution for totally 75 ml which divided by 25 ml inject into medial gutter and 25 ml inject into lateral gutter before cementation and implantation. And the last 25 ml of multimodal analgesic drugs were injected into quadriceps.

ELIGIBILITY:
Inclusion Criteria:

* 50 - 80 yrs of age ASA classification: 1-3 Unilateral TKA

Exclusion Criteria:

* Secondary OA knee Previous knee surgery Can't undertaken spinal block and adductor canal block Renal insuf. (Crcl < 30 ml/min) History of convulsive disorder Abnormal liver function BMI > 35 Kg/M2 Allergy to study drugs History of coronary disease Hb < 10 (g/dl) Can't understand 100mm-VAS assessment Refuse to recruit in the study, or refuse follow up Using opioid in 5 days before surgery Unstable vital sign History current VTE Using anti-platelet or anti-coagulation medicine Severe deformity

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
pain scores | at 4, 6 hours and every 6 hours after surgery for 2 days, then daily for 2 weeks after surgery.
  Visual analog scale at rest and motion (0-100 points, 0 mean best, 100 mean worst)

SECONDARY OUTCOMES:
Morphine consumption | 2 weeks
  Morphine consumption in hospital 48 hours before discharge and MST as home medication for 2 weeks (MME)
number of vomit events | at first 48 hours before discharge and after discharge for 2 weeks after surgery
  number of vomit events
Number of other Events of Morphine side effect | 2 weeks after surgery
  Itching, rash, constipation, difficult urination, respiratory, etc.
ROM | before surgery and 24, 48hours and 2 weeks after surgery
  ROM (degree)
Timed up and go test | at 48 hours and 2 weeks after surgery
  start with standing and then walk for 3 meters, then turn back to seat for 3 meters, then sit (report in seconds)
Length of stays in hospital | up to 72 hours
  Number of hours the patient stays for surgery
Time to walk | up to 48 hours
  hours after surgery of patients at first start walking to the toilet
Operative time | up to 2 hours
  duration from start incision to wound closure in TKA procedure (minutes)
Number of other complication | 2 weeks
  clinical VTE, wound and skin complication, superficial and deep infection

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University Hospital, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McNamara CA, Laurita J, Lambert BS, Sullivan TC, Clyburn TA, Incavo SJ, Park KJ. A multimodal intraosseous infusion of morphine and ketorolac decreases early postoperative pain and opioid consumption following total knee arthroplasty. Knee. 2023 Aug;43:129-135. doi: 10.1016/j.knee.2023.06.002. Epub 2023 Jul 1. PMID 37399631
- [Background] Lamplot JD, Wagner ER, Manning DW. Multimodal pain management in total knee arthroplasty: a prospective randomized controlled trial. J Arthroplasty. 2014 Feb;29(2):329-34. doi: 10.1016/j.arth.2013.06.005. Epub 2013 Jul 11. PMID 23850410
- [Background] Brozovich AA, Incavo SJ, Lambert BS, Sullivan TC, Wininger AE, Clyburn TA, Taraballi F, Park KJ. Intraosseous Morphine Decreases Postoperative Pain and Pain Medication Use in Total Knee Arthroplasty: A Double-Blind, Randomized Controlled Trial. J Arthroplasty. 2022 Jun;37(6S):S139-S146. doi: 10.1016/j.arth.2021.10.009. Epub 2022 Mar 7. PMID 35272897